CLINICAL TRIAL: NCT03624101
Title: Novel Therapeutic Approaches for Treatment of CF Patients With W1282X Premature Termination Codon Mutations
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: summary results revealed ineffective intervention and the trial was terminated prematurely. No formal statistical analysis was performed
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Steven M Rowe, Principal Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300001363
Record Dates: First submitted 2018-08-07; First posted 2018-08-09 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — tezacaftor, ivacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Symdeko (Experimental): If the participant is not on a current modulator, they will take Symdeko for 28 days followed by a 28 day off period. This cycle will be continued for 168 days
  Interventions: Drug: Symdeko
- Symdeko/Trikafta (Experimental): If the participant currently takes Symdeko , they will take Trikafta for a 28 day period followed by Symdeko for a 28 day period. This cycle will be continued for 168 days
  Interventions: Drug: Ivacaftor and Symdeko

INTERVENTIONS:
Drug: Symdeko — CFTR modulator
  Arms: Symdeko
Drug: Ivacaftor and Symdeko — CFTR modulator
  Arms: Symdeko/Trikafta

SUMMARY:
Based on previous clinical findings, the investigator hypothesize that ivacaftor will have synergistic effects with drugs that facilitate truncated but partially active W1282X CFTR protein processing (tezacaftor) in patients with W1282X CFTR. In the current study, the investigators propose to directly test the efficacy of tezacaftor/ivacaftor (TEZ/IVA) and Trikafta for W1282X CFTR therapy in the clinic in comparison to ivacaftor alone.

DETAILED DESCRIPTION:
Approximately 11% of CF patients have premature termination codons (PTC), causing truncated CFTR with little to no function. No approved therapies exist for patients with PTC mutations including W1282X, a unique mutation exhibiting partial CFTR activity even in its truncated form. CFTR modulators alone enhanced CFTR function in patient cells from W1282X/G542X CFTR. Several published studies have shown CFTR modulators alone and/or in combination with readthrough (RT) agents benefit W1282X CFTR. Clinical studies further support an aspect of this notion, where two W1282X patients showed beneficial effect to Ivacaftor treatment.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of signed and dated informed consent/assent document(s) indicating that the subject (and/or his parent/legal guardian) has been informed of all pertinent aspects of the trial

  * Age ≥ 18 yrs
  * Body weight ≥ 16 kg
  * Diagnosis of CF and documentation of the presence of a nonsense mutation of the CFTR gene, as determined by historical genotyping
  * Ability to perform a valid, reproducible spirometry with demonstration of FEV1 ≥ 30% and ≤ 90% of predicted for age, gender, and height
  * In subjects who are sexually active, willingness to abstain from sexual intercourse or employ a barrier or medical method of contraception during the study drug administration
  * Willingness and ability to comply with all study procedures and assessments

Exclusion Criteria:

* Any change (initiation, change in type of drug, dose modification, schedule modification, interruption, discontinuation, or re-initiation) in a chronic treatment/prophylaxis regimen for CF or for CF-related conditions within 2 weeks prior to screening
* Ongoing participation in any other therapeutic clinical trial
* Evidence of pulmonary exacerbation or acute upper or lower respiratory tract infection (including viral illnesses) within 2 weeks prior to screening
* History of solid organ or hematological transplantation; positive hepatitis B surface antigen test; hepatitis C antibody test; or human immunodecifiency
* Major complication of lung disease (including massive hemoptysis, pneumothorax, or pleural effusion) within 4 weeks prior to screening
* Pregnancy or breast-feeding
* Current smoker or a smoking history of ≥ 10 pack-years (number of cigarette packs/day x number of years smoked)
* Prior or ongoing medical condition (eg, renal failure, alcoholism, drug abuse, psychiatric condition), medical history, physical findings, ECG findings, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the subject, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Symdeko/Ivacaftor: If the participant currently takes Symdeko and Ivacaftor, they will take Symdeko for a 28 day period followed by Ivacaftor for a 28 day period. This cycle will be continued for 168 days
  symdeko/Ivacaftor: CFTR modulator
Period: Overall Study
Arm/Group | Symdeko | Symdeko/Ivacaftor
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: only 1 patient was enrolled into the study and was enrolled into the symdeko arm. No pateints were enrolled into the symdeko/ivacaftor arm
Groups:
- Symdeko: If the participant is on symdeko, they will take symdeko for 28 days followed by a 28 day off period. This cycle will be continued for 168 day
  Symdeko: CFTR modulator
- Symdeko/Ivacaftor: If the participant currently takes Symdeko , they will take Symdeko for a 28 day period followed by Ivacaftor for a 28 day period. This cycle will be continued for 168 days
  symdeko/Ivacaftor: CFTR modulator
- Total: Total of all reporting groups
Arm/Group | Symdeko | Symdeko/Ivacaftor | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 37 [37 to 37] |  | 37 [37 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in FEV1 From Baseline
Description: Percent change in FEV1 from Baseline and 24 weeks
Time Frame: 24 weeks
Population: no improvement was noticed and the study ended prematurely. No formal statistical analysis was performed
Measure: Number; unit: change in percentage
Groups:
- Symdeko/Ivacaftor: If the participant currently takes Symdeko, they will take Symdeko for a 28 day period followed by Ivacaftor for a 28 day period. This cycle will be continued for 168 days
  symdeko/Ivacaftor: CFTR modulator
Arm/Group | Symdeko | Symdeko/Ivacaftor
Number analyzed (Participants) | 1 | 0
change in percentage | 0 |

ADVERSE EVENTS:
Time Frame: 6 months
Description: only 1 patient was entered into the study (Symdeko Arm). No patients were entered into the Symdeko/Ivacaftor Arm
Arm/Group | Symdeko | Symdeko/Ivacaftor
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Symdeko (N=1) | Symdeko/Ivacaftor (N=0)
Increased cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
increased sputum production (Respiratory, thoracic and mediastinal disorders) | 1 (2) | NA
Increased fatigue (General disorders) | 1 (2) | NA
decreased appetite (Metabolism and nutrition disorders) | 1 (1) | NA
low blood glucose (Endocrine disorders) | 1 (1) | NA

LIMITATIONS AND CAVEATS:
the data collected was not compelling enough to move forward and no publications or official findings were available

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-19): https://cdn.clinicaltrials.gov/large-docs/01/NCT03624101/Prot_SAP_000.pdf